CLINICAL TRIAL: NCT05104216
Title: Immunogenicity and Safety of a Third Dose and Immune Persistence of BBIBP-Corv Vaccine in Elderly People With Chronic Bronchitis and Chronic Obstructive Pulmonary Disease
Brief Title: Immunogenicity and Safety of a Third Dose and Immune Persistence of BBIBP-Corv Vaccine in Elderly People With Chronic Bronchitis and COPD
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: China National Biotec Group Company Limited (Industry)
Collaborators: Zhejiang Provincial Center for Disease Control and Prevention (Other Government); Beijing Institute of Biological Products Co Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: BIBP2021COPD-third dose
Record Dates: First submitted 2021-10-21; First posted 2021-11-02 (Actual); Last update posted 2021-11-02 (Actual); Status verified 2021-10

CONDITIONS: COVID-19; Chronic Bronchitis; COPD
MeSH Terms: conditions — COVID-19; Bronchitis, Chronic; Pulmonary Disease, Chronic Obstructive

STUDY DESIGN:
Intervention Model Description: Subjects aged ≥60 with chronic bronchitis and COPD who have completed the schedule of two doses for 3 months receive a third dose of inactivated COVID-19 vaccine.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Experimental Group (Experimental): Subjects receive a third dose of inactivated COVID-19 vaccine
  Interventions: Biological: Inactivated COVID-19 vaccine

INTERVENTIONS:
Biological: Inactivated COVID-19 vaccine — receive a third dose of inactivated COVID-19 vaccine

SUMMARY:
Evaluation of immunogenicity, safety and persistence of the subjects aged 60 years and above with chronic bronchitis and chronic obstructive pulmonary disease received the third dose of inactivated COVID-19 vaccine .

DETAILED DESCRIPTION:
The subjects aged 60 years and above with chronic bronchitis and chronic obstructive pulmonary disease recruited to receive a third dose of inactivated COVID-19 vaccine.

Blood samples will be collected 3 times: before the third dose of vaccinatioin，28 days and 6 months after the third dose of vaccination.

Any local or systemic adverse events that occurred within 21 days after vaccination will be recorded.

ELIGIBILITY:
Inclusion Criteria:

* Subjects aged 60 and above with full capacity for civil conduct;
* Chronic bronchitis (or chronic obstructive pulmonary disease) diagnosed by a medical institution at level I or above;
* Body temperature < 37.3 ° C confirmed by clinical examination before enrollment ;
* Able and willing to complete the entire study plan during the study follow-up period;
* Have the ability to understand the study procedures, voluntarily sign informed consent, and comply with the requirements of the clinical study protocol;
* Subjects participating in the past clinical trial have completed two doses of COVID-19 vaccine and blood collection before and after immunization;

Exclusion Criteria:

* Subjects were previously confirmed cases of COVID-19 or asymptomatic infected persons;
* Being allergic to any component of vaccines (including excipients) ;
* Injection of non-specific immunoglobulin within 1 month before enrollment;
* Injection of live attenuated vaccines within 1 month and injection of other vaccines within 14 days before enrollment;
* Subjects who have experienced severe allergic reactions to vaccines (e.g. acute anaphylaxis, urticaria, angioneurotic edema, dyspnea, etc.);
* Having uncontrolled epilepsy and other progressive neurological disorders and a history of Guillain-Barre syndrome;
* Having severe liver and kidney diseases, malignant tumors, acute diseases or acute episodes of chronic diseases;
* Have been diagnosed with congenital or acquired immunodeficiency, HIV infection, lymphoma, leukaemia or other autoimmune diseases;
* Have been diagnosed with thrombocytopenia or other clotting disorders that may contraindicate subcutaneous injection;
* During an acute episode of chronic bronchitis/chronic obstructive pulmonary disease;
* Subjects who had vaccine-related adverse reactions after the second dose;
* Having high fever (axillary temperature ≥39.0℃) for three days after the second dose of inoculation, or severe allergic reaction;
* Having any adverse nervous system reaction after the second dose;
* During the acute onset of a chronic disease, or the recovery of acute complications less than two weeks;
* Other reasons for exclusion considered by the investigator.

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 400 (Estimated)
Dates: Start 2021-12 (Estimated); Primary Completion 2022-06-30 (Estimated); Study Completion 2022-06-30 (Estimated)

PRIMARY OUTCOMES:
Seroconversion rate | 28 days after the 3th dose (Day 28)
  The rate of seroconversion against coronavirus
Neutralizing antibody level | Before the 3th dose (Day 0)
  Neutralizing antibody GMT against coronavirus before the 3th dose
Neutralizing antibody level | 28 days after the 3th dose (Day 28)
  Neutralizing antibody GMT against coronavirus after the 3th dose
Neutralizing antibody level | 6 months after the 3th dose
  Neutralizing antibody GMT against coronavirus after the 3th dose

SECONDARY OUTCOMES:
Adverse events rate | 0-21days following vaccinations
  Analyse the incidence of adverse events following vaccination, both solicited and unsolicited
Serious adverse event rate | 0-6 months
  Report and analyse serious adverse events

CONTACTS AND LOCATIONS:
Overall Officials: Hanqing He, Principal Investigator — Zhejiang Provincial Center for Disease Control and Prevention
Locations (1):
- Zhejiang provincial center for disease control and prevention, Hangzhou, Zhejiang, China